CLINICAL TRIAL: NCT00333502
Title: A Phase 1b/2a Safety and Pharmacokinetic Study of CRLX101 (Formerly Named IT-101) in the Treatment of Advanced Solid Tumors
Brief Title: Study of CRLX101 (NLG207) in the Treatment of Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRLX-001; City of Hope IRB number 05127
Record Dates: First submitted 2006-06-01; First posted 2006-06-05 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Cancer; Solid Tumor
Keywords: Cancer, Neoplasms, Solid Tumor, Ovarian Cancer, Lung Cancer,; Non Small Cell Lung Cancer, Pancreatic Cancer,; Breast Cancer, Colon Cancer, Endometrial Cancer,; Kidney (Renal Cell) Cancer, Melanoma, Prostate Cancer,; Skin Cancer, Thyroid Cancer,; Solid Malignancies
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Breast Neoplasms; Colonic Neoplasms; Endometrial Neoplasms; Melanoma; Prostatic Neoplasms; Skin Neoplasms; Thyroid Neoplasms | interventions — Camptothecin; 2-cyclohexylidenhydrazo-4-phenyl-thiazole; IT-101

ARMS (1):
- CRLX101 (formerly known as IT-101) (Experimental): CRLX101 dosing per protocol dose escalation cohorts to MTD, then expansion cohort treated at MTD of CRLX101 15mg/m2
  Interventions: Drug: Camptothecin (CPT) conjugated to a linear, cyclodextrin-based polymer

INTERVENTIONS:
Drug: Camptothecin (CPT) conjugated to a linear, cyclodextrin-based polymer — Subjects who meet inclusion/exclusion criteria will receive CRLX101 every other week.
  Other Names: NLG207; IT-101

SUMMARY:
CRLX101 is a nanopharmaceutical comprised of the chemotherapeutic camptothecin (CPT) conjugated to a linear, cyclodextrin-based polymer. CRLX101 is designed to increase the exposure of tumor cells to CPT while minimizing side effects.

OBJECTIVES:

• Determine the safety, toxicity, and the maximum tolerated dose (MTD) of CRLX101 when administered intravenously to subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects >18 years of age with advanced, histologically-confirmed solid tumors refractory to standard therapy or for which no standard therapy exists and who have evidence of disease progression documented since their prior therapy.
* Subjects must have measurable or evaluable disease.
* Subjects must not have received prior chemotherapy or radiation for >/= 4 weeks prior to first dose of study drug.
* Subjects may be entered if they have received prior radiation therapy involving </= 30% of the bone marrow. Any prior radiation therapy must have been administered >/= 4 weeks prior to first dose of study drug and the subject must be recovered from the acute toxic effects of the treatment prior to study entry.
* Subjects may be enrolled with a history of treated brain metastases that are clinically stable for >/= 4 weeks prior to first dose of study drug. Subjects may not be currently receiving dexamethasone.
* ECOG performance status of < 2.
* Life expectancy of greater than 12 weeks.
* Subjects must have acceptable organ and marrow function at screening and pre-dose visits.
* Electrocardiogram without evidence of clinically significant conduction abnormalities or active ischemia as determined by the investigator and an acceptable QTc interval.
* The effects of CRLX101 on the developing human fetus are unknown, therefore, women of childbearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Female subjects who are pregnant or nursing.
* Subjects who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to first dose of study drug or those who have not had adverse events return to baseline severity level or a severity level Grade 1 due to agents administered more than 4 weeks prior to first dose of study drug.
* Subjects with a history of congestive heart failure (CHF) requiring medical therapy.
* Subjects with serum amylase or lipase > 1.5X upper limit of normal (ULN).
* Subjects with previous high dose chemotherapy with autologous stem cell rescue bone marrow transplantation.
* Use of any investigational agent or drug within 4 weeks prior to first dose of study drug.
* Metastatic disease to the CNS requiring treatment or radiation therapy.
* Subjects with known untreated brain metastases or treated brain metastases that have not been stable >/= 4 weeks prior to first dose of study drug.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, hypertension, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, as determined by the investigator.
* The presence of active coagulation disorder.
* Subjects with marked baseline prolongation of QT/QTc interval (QTc interval >/= 470 msec for females and QTc interval >/= 450 msec for males).
* Any prior treatment with a topoisomerase I inhibitor.
* Any major surgery </= 4 weeks prior to first dose of study drug.
* Concurrent use of G-CSF or growth factors at the time of initiation of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-05; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety, toxicity and maximum tolerated dose of CRLX101 when administered intravenously to subjects with advanced solid tumors. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yun Yen, M.D., Ph.D., Principal Investigator — City of Hope National Medical Center; Glenn Weiss, M.D., Principal Investigator — Virginia G. Piper Cancer Center; Jeffrey D. Neidhart, M.D., Principal Investigator — San Juan Oncology Associates
Locations (3):
- United States (3):
  - Virginia G. Piper Cancer Center, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - San Juan Oncology Associates, Farmington, New Mexico

REFERENCES:
- [Background] Schluep T, Hwang J, Cheng J, Heidel JD, Bartlett DW, Hollister B, Davis ME. Preclinical efficacy of the camptothecin-polymer conjugate IT-101 in multiple cancer models. Clin Cancer Res. 2006 Mar 1;12(5):1606-14. doi: 10.1158/1078-0432.CCR-05-1566. PMID 16533788
- [Background] Schluep T, Cheng J, Khin KT, Davis ME. Pharmacokinetics and biodistribution of the camptothecin-polymer conjugate IT-101 in rats and tumor-bearing mice. Cancer Chemother Pharmacol. 2006 May;57(5):654-62. doi: 10.1007/s00280-005-0091-7. Epub 2005 Aug 26. PMID 16133526
- [Background] Cheng J, Khin KT, Davis ME. Antitumor activity of beta-cyclodextrin polymer-camptothecin conjugates. Mol Pharm. 2004 May-Jun;1(3):183-93. doi: 10.1021/mp049966y. PMID 15981921